CLINICAL TRIAL: NCT04459078
Title: A Prospective Single-arm Phase II Clinical Study to Evaluate the Efficacy of Camrelizumab in Combined With APatinib and Albumin Paclitacxel in Advanced Untreated EGFR Wild Type and ALK-negative Lung Adenocarcinoma
Brief Title: Clinical Study of Camrelizumab Combined With APatinib and Albumin Paclitacxel in Patients With Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Suzhou Sheng Diya Biomedical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Lin Wu, Chief physician, director of department, Hunan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPAP-lung
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Adenocarcinoma of the Lung
Keywords: immunotherapy; PD-1 checkpoint inhibitor; Anti-angiogenesis; First-line Treatment
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — camrelizumab; Immune Checkpoint Inhibitors; apatinib; Angiogenesis Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be enrolled into our study. Participants are given intravenous administration of Camrelizumab (200mg/3w) in addition with intravenous administration of Albumin Paclitacxel (135mg/m2, d1, d8/3w, 4-6 cycles) and Apatinib (250mg Qd po for 5 days, take rest for 2 days every week). Treatment terminates when disease progression, death or unacceptable toxicity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with Albumin Paclitacxel and Apatinib. (Experimental): Participants are given intravenous administration of Camrelizumab (200mg/3w) in addition with intravenous administration of Albumin Paclitacxel (135mg/m2, d1, d8/3w, 4-6 cycles) and Apatinib (250mg Qd po for 5 days,, take rest for 2 days every week). Treatment terminates when disease progression, death or unacceptable toxicity.
  Interventions: Drug: Camrelizumab; Drug: Albumin Paclitacxel; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Intravenous administration of (200mg/3weeks)
  Other Names: SHR1210; PD-1 inhibitor
Drug: Albumin Paclitacxel — intravenous administration of Albumin Paclitacxel (135mg/m2, d1, d8/3w, 4-6 cycles)
  Other Names: Chemotherapy drug
Drug: Apatinib — Patients will be given oral of Apatinib (250mg Qd po for 5 days, take rest for 2 days every week)
  Other Names: Anti-angiogenesis drug

SUMMARY:
This study is a single arm, open label, national multicenter study, to explore the efficacy and safety of the combination of Camrelizumab, apatinib and albumin paclitaxel in advanced untreated EGFR Wild Type and ALK-negative Lung Adenocarcinoma. The study does not consider PD-L1 expression, but tumor samples need to be explored by PD-L1 detection and other exploratory analysis.

DETAILED DESCRIPTION:
Primary outcome:

1. progression free survival (PFS) evaluated according to RECIST1.1.

Secondary outcome:

1. Objective Response Rate (ORR), Overall Survival (OS), Disease Control Rate (DCR), Duration of Response (DOR) evaluated according to RECIST1.1, and Quality of Life(QOL).
2. The overall incidence of adverse events (AE); the incidence of grade 3 or above AE; the incidence of serious adverse events (SAE); the incidence of AE leading to the termination of the trial drug; the incidence of AE leading to the suspension of the trial drug.
3. Exploratory analysis of potential biomarkers related to efficacy. The characteristics of tumor tissue PD-L1expression, panel-captured next generation sequencing(NGS), RNA-seq, T-Cell Repertoire (TCR), multiple immunofluorescence and other biomarkers, and the correlation analysis of biomarkers with efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age>=18 years, both men and women can be enrolled 2. Histologically confirmed adenocarcinoma (does not contain small cell components).

  3. Locally advanced, untreated recurrent or metastatic lung adenocarcinoma not suitable for radical surgery or radiotherapy. Previous neoadjuvant and adjuvant radiochemotherapy can be accepted (chemotherapy/radiotherapy, non-immunotherapy), tumor progression ≥6 months before the end of neoadjuvant / adjuvant therapy is required .

  4. ECOG score of physical condition was 0-1, and there was no deterioration in the first 2 weeks. Expected survival over 12 weeks.

  5. According to the RECIST1.1 criteria, it is required that at least one measurable treatment naive lesion (has not been treated with radiotherapy in the past and will not receive local therapy such as radiotherapy throughout the treatment); If the lesion has been treated with radiotherapy then the progress of this lesion need to be confirmed by imaging, before being used as the target lesion.

  6. Laboratory certified by CAP reported negative in EGFR and ALK mutation-sensitive mutations.

  7. Clinical laboratory examination indicators meet the following standards:
  1. Platelet ≥100×109/L
  2. Absolute neutrophil count (ANC) ≥1.5×109/L, or absolute white blood cell count (WBC) ≥3.5×109/L
  3. Hemoglobin (Hgb) ≥ 100 g/L (without blood transfusion or erythropoietin use within 4 weeks)
  4. Total bilirubin ≤ 1.5 times the upper limit of normal value (ULN) (If there is liver metastasis, allow ≤2.5 times ULN)
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN
  6. Creatinine ≤1.5 times ULN or Creatinine clearance ≥50 mL/min (Calculated according to the Cockcroft Gault formula)
  7. Serum amylase ≤ 2 times ULN or pancreatic amylase ≤ 1.5 times ULN
  8. Serum lipase ≤ 1.5 times ULN
  9. patients who did not take anticoagulants, or those who had previously used anticoagulants, had been discontinued for 28 days before enrollment, and the international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.

     8. Able to swallow oral medication. 9. Enough tissue specimens for PD-L1 detection or exploratory analysis.

     Exclusion Criteria:
* 1.The histological component of NSCLC containing small cell lung cancer or squamous cell carcinoma was excluded.

  2. Previously untreated or symptomatic central nervous system (CNS) metastases or meningeal diseases, spinal cord compression, meningeal metastases and brain metastases with obvious symptoms, etc. For those who have received radiotherapy and/or surgery, patients with no evidence of CNS disease progression ≥ 2 weeks after the end of treatment, patients who had not been treated with corticosteroids for more than 2 weeks before the start of treatment were eligible.

  3. Clinically significant hemoptysis (at least 0.5 teaspoons of fresh blood) or tumor bleeding occurred within 2 weeks before the first dose of study treatment.

  4. There is imaging evidence of invasion/infiltration of large vessels. Due to the potential risk of severe bleeding associated with tumor shrinkage/necrosis after apatinib treatment, the degree of tumor invasion/infiltration of major blood vessels should be considered.

  5. Cancerous thrombus with clinical significance, and the use of anticoagulant drugs within 28 days before enrollment.

  6. Clinically uncontrollable pleural effusion/abdominal effusion. 7. Glucocorticoid treatment 28 days before the first dose (equivalent dose of >10 mg prednisone per day).

  8. Having active autoimmune diseases, which require systemic treatment in the past 2 years (ie using disease-modifying drugs, corticosteroids or immunosuppressive drugs). Replacement therapy (for example, thyroxine, insulin, or physiological corticosteroid replacement therapy due to adrenal or pituitary insufficiency, etc.) is not considered as systemic therapy and is allowed.

  9. History of other malignant tumors in the past 5 years. 10. Has received previous systemic chemotherapy or other targeted or biological anti-tumor treatment for its metastatic NSCLC (As long as treatment is completed at least 6 months before diagnosis of metastatic NSCLC, prior chemotherapy and/or radiotherapy is allowed as part of neoadjuvant/adjuvant therapy for non-metastatic NSCLC).

  11. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2 and other drugs or drugs acting on another stimulatory or co-suppressive T cell receptor (eg CTLA-4, OX 40, CD137 ) therapy, or cell biological therapy, etc.

  12. Previously received treatment with apatinib, or received systemic medication with a clear anti-tumor mechanism.

  13. Allogeneic tissue/solid organ transplantation has been performed. 14. In addition to hair loss and stable peripheral neurotoxicity below grade 2, any clinical toxicity associated with prior treatment before enrollment did not return to pre-treatment levels or grade 1.

  15. pregnancy status (positive blood HCG) and lactation. 16. Previously suffering from interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring hormone therapy, or any active interstitial lung disease with clinical evidence.

  17. Known liver diseases of clinical significance, including active viral hepatitis, alcoholic hepatitis or other hepatitis, liver cirrhosis, hereditary liver disease.( patients who have been cured of previous HBV infection (defined as hepatitis B core antibody [HBcAb] positive and HBsAg negative) can participate in this study. Before entering the group, HBV DNA testing must be performed on this class of patients and well-controlled hepatitis B (peripheral HBV DNA testing is less than 103/ml) can be considered for this experiment, and antiviral treatment should be given. Previous patients infected with hepatitis C virus (HCV) had positive HCV antibody test results, They were eligible for this study only if the HCV RNA polymerase chain reaction test result was negative (below the detection limit).) 18. Patients who are suspected or have demonstrated an impaired immune function or infection, including:
  * Evidence that active or latent tuberculosis (TB) is determined by locally approved screening methods. If the screening results require treatment in accordance with local treatment guidelines or clinical practice, the patient is disqualified.
  * Chronic or active hepatitis B or hepatitis C.
  * Known history of human immunodeficiency virus (HIV) infection. During the screening period, the local test result was positive.
  * There are any other medical conditions (such as active infections that have been treated or not treated) that the investigator believes that the patient has an unacceptable risk if receiving immunomodulatory therapy(Patients with local diseases that are unlikely to cause systemic infections (such as chronic nail fungal infections) are allowed to be enrolled).

    19. Allogeneic bone marrow or organ transplantation. 20. Any immunomodulator with systemic effects. 21. Known mental illness or substance abuse disorders that interfere with a subject's ability to comply with research requirements.

    22. Previous severe allergy to mAb treatment or known allergy or intolerance to any component of study medication (apatinib, caririzumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 24 months
  Progression free survival (PFS) evaluated by investigators based on the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
ORR | Up to 24 months
  Objective Remission Rate (ORR) evaluated by researchers based on the RECIST 1.1 criteria.
OS | Up to 24 months
  Overall Survival (OS) evaluated by researchers based on the RECIST 1.1 criteria.
DCR | Up to 24 months
  Disease Control Rate（DCR）evaluated by researchers based on the RECIST 1.1 criteria.
DOR | Up to 24 months
  Duration of Response (DOR) evaluated by researchers based on the RECIST 1.1 criteria.
The change of quality of life | Up to 24 months
  The change of quality of life is measured using the European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnaire（EORTC QLQ）
AE | Up to 24 months
  The overall incidence of adverse events (AE); the incidence of grade 3 or above AE; the incidence of serious adverse events (SAE); the incidence of AE leading to the termination of the trial drug; the incidence of AE leading to the suspension of the trial drug

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Hunan Cancer hospital, Changsha, Hunan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work.

REFERENCES:
- [Derived] Pu X, Lin G, Xiao M, Lin J, Wang Q, Kong Y, Yan X, Xu F, Xu Y, Li J, Li K, Chen B, Wen X, Tan Y, Cheng F, Zhu K, Li N, Wu L. Camrelizumab combined with apatinib and nanoparticle albumin-bound paclitaxel in lung adenocarcinoma (CAPAP-lung): a single-arm phase II study. EClinicalMedicine. 2024 Jan 3;67:102403. doi: 10.1016/j.eclinm.2023.102403. eCollection 2024 Jan. PMID 38261958